CLINICAL TRIAL: NCT01752803
Title: A Double-blind, Randomized Placebo-controlled Parallel Group Study of Probiotics as an Adjuvant Therapy for Individuals With Type 2 Diabetes Mellitus
Brief Title: RCT Examining Effects of Probiotics in T2DM Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-02-12-1815RU; Universiti Putra Malaysia (Other Grant/Funding Number: Universiti Putra Malaysia)
Record Dates: First submitted 2012-12-16; First posted 2012-12-19 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes Mellitus; Obesity; Hypertension; Hyperlipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Hypertension; Hyperlipidemias | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotic (Experimental): subjects in this arm will receive probiotic supplementation for 12 weeks.
  Interventions: Dietary Supplement: Probiotic
- placebo (Placebo Comparator): subjects in this arm will receive placebo in identical sachets similar to probiotics which only differs in the codes mentioned on the label of sachets.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — mix probiotic
  Other Names: mix probiotic supplementation
  Arms: probiotic
Dietary Supplement: Placebo — placebo
  Arms: placebo

SUMMARY:
Background: The connection between gut health and diabetes status is increasingly recognized. Gut microbiota composition in diabetic differs from non-diabetic individuals. Interestingly, the level of glucose tolerance was associated with specific microbiota that was rarely found in healthy individuals. Probiotics is one of the functional foods believed to mediate their health promoting activities through modulating the composition of the gut health. Ingestion of probiotics has been shown not only to influence gut microbiota composition but also the secretion of the gut hormones and insulin resistance in animal models with limited trials in human. Supplementation with probiotic has also been shown not only affect glucose homeostasis, but improved other diabetes related comorbidities such as obesity, hypertension, and hyperlipidemia.

Objectives and hypotheses: To address this research gap, this Randomized Controlled Trial (RCT) is proposed to determine the efficacy of probiotic supplementations as adjuvant therapy to improve glucose homeostasis through modulating gut microbiota composition and gut hormones secretion in individuals with type 2 diabetes. We hypothesized that the probiotic supplementations will improve blood glucose control as well as other diabetes related co-morbidities in individuals with type 2 diabetes.

Methodology: This is a double blind randomized parallel group control trial with 3 months probiotic supplementation or placebo. After screening the eligible subjects will be selected. Then, after consent taking, subjects will be randomly assigned to either receive probiotic or supplement for 3 months. Measurements of blood parameters including glycemic control related parameters, lipid profile, renal profile, and liver function tests as well as three day diet recall, and anthropometry measurements will take place at baseline, after 6 weeks and after 12 months.

Expected Outcomes: Probiotic supplementation as an adjuvant therapy would improve glucose homeostasis and gut health as compared to the placebo and eventually will beneficially affect other diabetes related conditions. This study would provide avenue to identify the possibility of probiotic supplementations as an adjuvant therapy in the management of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Established type 2 diabetes with at least 6 months diagnosis
2. Age between 30 and 65 years
3. Hb A1c of less than 10% and fasting blood glucose less than 15mmol/l
4. BMI between 18.5-35 kg/ m2
5. Have not on any probiotics for the last 2 months prior to the recruitment
6. Ability to comply to the study protocol
7. They are treated with stabilized dose of medications (either receiving Sulphonylurea or Biguanides or both)

Exclusion Criteria:

1. Pregnancy and lactating (subjects will be excluded if they getting pregnant during course of study)
2. Having advanced diabetes complications except for hypertension and hyperlipidemia
3. Having acute or chronic illness (such as flu, cancer or arthritis rheumatoid) during the study recruitment which may affect carbohydrate metabolism
4. Language barriers which cannot be overcome via available resources
5. Currently being treated with any oral anti-diabetes agents other than Sulphonylurea or Biguanides or being treated with insulin
6. Using any medication such as steroids or antibiotics which might affect viability of gut microorganism at recruitment and during intervention phase.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Hb A1c | 3 months

SECONDARY OUTCOMES:
inflammatory markers | 3 months

OTHER OUTCOMES:
Lipoproteins | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Somayyeh Firouzi, Master, Principal Investigator — Nutrition and Dietetic department, University Putra Malaysia
Locations (1):
- Universiti Kebangsaan Malaysia Medical Center, Kuala Lumpur, WP, Malaysia

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148
- [Derived] Firouzi S, Mohd-Yusof BN, Majid HA, Ismail A, Kamaruddin NA. Effect of microbial cell preparation on renal profile and liver function among type 2 diabetics: a randomized controlled trial. BMC Complement Altern Med. 2015 Dec 12;15:433. doi: 10.1186/s12906-015-0952-5. PMID 26654906